CLINICAL TRIAL: NCT04552236
Title: Evaluation of Liver Stiffness by Ultrasound Elastography for Predicting Early Hepatocellular Carcinoma Recurrence After Treatment
Brief Title: Evaluation of Liver Stiffness by Ultrasound Elastography for Predicting Early HCC Recurrence After Treatment
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Reem Mohamed Saad EL Shazly, Principle investigator, Assiut University
Other Study IDs: Ultrasound Elastography in HCC
Record Dates: First submitted 2020-09-11; First posted 2020-09-17 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Ultrasound ELastography — A standardized liver Elastography is critical to obtain reliable and accurate results . The patient is imaged in supine or slight 30 degrees left lateral decubitus position, with the right arm elevated above the head to open the intercostal spaces and improve the acoustic window to the liver . it is recommended to sample measurements in the right lobe , which has shown the most reliable results. Transducer pressure on the skin should be similar to regular anatomical B-mode imaging.
  When using SWE techniques, the acoustic radiation force push pulse should be applied perpendicular to the liver capsule, with measurements obtained 4-5 cm deep to the skin and within a minimum 1-2 cm of liver parenchyma to limit refraction of the pulse. The operator should verify that these areas are free of vascular and biliary structures and rib shadows.

SUMMARY:
We aim to evaluate liver stiffness as a marker of severity and duration of the underlying liver disease to predict for early HCC recurrence after treatment.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is one of the most common cancers worldwide and contributes to enormous cancer-related deaths annually . Hepatocellular carcinoma is a frequent complication of liver disease. Early recurrence is mainly tumour or treatment-related .

Liver fibrosis stagging is essential to evaluate the expected prognosis against the concomitant therapies. Liver biopsy remain the gold standard for diagnosing liver fibrosis, however, it is limited due to the associated costs, invasiveness, and intra and inter observer variability. Patient discomfort, refusal and risk of complications. Ultrasound Elastography is a non-invasive imaging method liver fibrosis staging . Ultrasound Elastography is an imaging technology sensitive to tissue stiffness that was developed in the 1990s. It has been further developed and refined in recent years to enable quantitative assessment of tissue stiffness. Elastography methods take advantage of the changed elasticity of soft tissues resulting from specific pathological or physiological processes .

Elastography is an application, which produces the force coupled with a measurement system for the deformities caused by the force. There are several types of forces: 1. static compression induced externally by manual compression or internally by organ motion (heart, vessel, and breathing) 2. Dynamic compression induced with a continuous vibration at a given frequency 3. Impulse compression (transient vibration) induced externally by a transient mechanical impulse ( Fibroscan) or internally by an ultrasound impulse (ARFI, SWE), both compression types producing shear waves. While contrast-enhanced imaging is the first-line approach in the diagnosis of HCC, recent report show that the non-invasively measured stiffness of hepatic nodule could help to distinguish between malignant and benign liver lesions.

The treatment of HCC depends on the stage of liver disease and in many cases, curative resection is not possible. Therefore local ablative therapies, such as transarterial chemoembolization (TACE) and radiofrequency ablation (RFA), are considered viable therapeutic options . However, HCC might behave very differently and could show more or less of a response to local ablative treatment

ELIGIBILITY:
Inclusion Criteria:

* All patients with liver cirrhosis and HCC.

Exclusion Criteria:

* Metastatic hepatic focal lesions.

Ages: 50 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with HCC and liver cirrhosis expected to visit Assiut university hospital to be treated
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Predicting early HCC recurrence after treatment by Ultrasound elastography | Baseline
  TO enhance surveillance and detect HCC recurrence as early as possible for further management

REFERENCES:
- [Background] Villanueva A. Hepatocellular Carcinoma. N Engl J Med. 2019 Apr 11;380(15):1450-1462. doi: 10.1056/NEJMra1713263. No abstract available. PMID 30970190
- [Background] Marasco G, Colecchia A, Colli A, Ravaioli F, Casazza G, Bacchi Reggiani ML, Cucchetti A, Cescon M, Festi D. Role of liver and spleen stiffness in predicting the recurrence of hepatocellular carcinoma after resection. J Hepatol. 2019 Mar;70(3):440-448. doi: 10.1016/j.jhep.2018.10.022. Epub 2018 Oct 31. PMID 30389551
- [Background] Attia D, Bantel H, Lenzen H, Manns MP, Gebel MJ, Potthoff A. Liver stiffness measurement using acoustic radiation force impulse elastography in overweight and obese patients. Aliment Pharmacol Ther. 2016 Aug;44(4):366-79. doi: 10.1111/apt.13710. Epub 2016 Jun 30. PMID 27363528
- [Background] Gennisson JL, Deffieux T, Fink M, Tanter M. Ultrasound elastography: principles and techniques. Diagn Interv Imaging. 2013 May;94(5):487-95. doi: 10.1016/j.diii.2013.01.022. Epub 2013 Apr 22. PMID 23619292
- [Background] Shiina T, Nightingale KR, Palmeri ML, Hall TJ, Bamber JC, Barr RG, Castera L, Choi BI, Chou YH, Cosgrove D, Dietrich CF, Ding H, Amy D, Farrokh A, Ferraioli G, Filice C, Friedrich-Rust M, Nakashima K, Schafer F, Sporea I, Suzuki S, Wilson S, Kudo M. WFUMB guidelines and recommendations for clinical use of ultrasound elastography: Part 1: basic principles and terminology. Ultrasound Med Biol. 2015 May;41(5):1126-47. doi: 10.1016/j.ultrasmedbio.2015.03.009. Epub 2015 Mar 21. PMID 25805059
- [Background] Roulot D, Czernichow S, Le Clesiau H, Costes JL, Vergnaud AC, Beaugrand M. Liver stiffness values in apparently healthy subjects: influence of gender and metabolic syndrome. J Hepatol. 2008 Apr;48(4):606-13. doi: 10.1016/j.jhep.2007.11.020. Epub 2008 Jan 3. PMID 18222014
- [Background] Jiao Y, Dong F, Wang H, Zhang L, Xu J, Zheng J, Fan H, Gan H, Chen L, Li M. Shear wave elastography imaging for detecting malignant lesions of the liver: a systematic review and pooled meta-analysis. Med Ultrason. 2017 Jan 31;19(1):16-22. doi: 10.11152/mu-925. PMID 28180192
- [Background] Conti CB, Cavalcoli F, Fraquelli M, Conte D, Massironi S. Ultrasound elastographic techniques in focal liver lesions. World J Gastroenterol. 2016 Mar 7;22(9):2647-56. doi: 10.3748/wjg.v22.i9.2647. PMID 26973405
- [Background] Grgurevic I, Bokun T, Salkic NN, Brkljacic B, Vukelic-Markovic M, Stoos-Veic T, Aralica G, Rakic M, Filipec-Kanizaj T, Berzigotti A. Liver elastography malignancy prediction score for noninvasive characterization of focal liver lesions. Liver Int. 2018 Jun;38(6):1055-1063. doi: 10.1111/liv.13611. Epub 2017 Nov 3. PMID 29028279
- [Background] European Association For The Study Of The Liver; European Organisation For Research And Treatment Of Cancer. EASL-EORTC clinical practice guidelines: management of hepatocellular carcinoma. J Hepatol. 2012 Apr;56(4):908-43. doi: 10.1016/j.jhep.2011.12.001. No abstract available. PMID 22424438
- [Background] Ho DWH, Chan LK, Chiu YT, Xu IMJ, Poon RTP, Cheung TT, Tang CN, Tang VWL, Lo ILO, Lam PWY, Yau DTW, Li MX, Wong CM, Ng IOL. TSC1/2 mutations define a molecular subset of HCC with aggressive behaviour and treatment implication. Gut. 2017 Aug;66(8):1496-1506. doi: 10.1136/gutjnl-2016-312734. Epub 2016 Dec 14. PMID 27974549
- Available data/document: Study Protocol — https://pubmed.ncbi.nlm.nih.gov/